CLINICAL TRIAL: NCT05214157
Title: A Prospective Randomized Controlled Study on the Role of Restoring Liver-Diaphragm Surface Tension and Pain Control at Port Sites in Optimizing Pain Management Following Laparoscopic Cholecystectomy
Brief Title: Optimizing Pain Management Following Laparoscopic Cholecystectomy RCT
Acronym: Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Mohamed lotfy, Associate professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: zuh 243
Record Dates: First submitted 2022-01-25; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Acute Post-operative Pain; Cholecystectomy, Laparoscopic; Pain Assessment Pain Intensity; Pain Intensity
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): interventional group, final two operative steps applied
  Interventions: Procedure: active gas aspiration
- group B (No Intervention): control group

INTERVENTIONS:
Procedure: active gas aspiration — sucking remaining Co2 from the peritoneal cavity and local anaesthetic application at port sites
  Other Names: application of Bupivacaine soaked sponge
  Arms: group A

SUMMARY:
evaluating the two final steps we added to optimize post laparoscopic cholecystectomy pain management.

DETAILED DESCRIPTION:
Introduction: After a laparoscopic cholecystectomy (LC), pain is still a significant concern, leading to extended hospital stays or readmissions. In majority of patients, postoperative pain medications are required. A standardized strategy is needed to offer effective pain relief postoperatively. The majority of pain in the early postoperative period is due to elimination of intraperitoneal surface tension or of parietal type. Aim of the work: to evaluate the two final steps we added to optimize postoperative pain management. Patients and methods: Over the period from March 2020 to December 2021, 816 patients with gallbladder stone undergoing LC were randomized into 2 groups after exclusion of 12 patients: Group A; interventional contained 402 patients. Group B; control contained 402 patients. Post-operative data to be compared were made in terms of operative time, shoulder pain, upper abdominal pain, (at 6,12,18 and 24 hours) and number of analgesic doses and hospital stay. Pain intensity was assessed by using the visual analogue scale (VAS) for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were having symptoms consistent with biliary colic,
* had ultrasound evidence of gall stones,
* classified as American Society of Anesthesiology (ASA) I and II
* ages ranging from 18 to 65 years

Exclusion Criteria:

* Patients who refused to give consent,
* pregnant,
* had a history of drug abuse,
* had CBD stones,
* acute cholecystitis,
* acute pancreatitis,
* previous abdominal surgery,
* history of peritonitis,
* had carcinoma of the gall bladder Patients who were converted to open surgery,
* patients who required placement of drains
* patients with intraoperative complications (CBD injury or liver bed bleeding).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 804 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-08 (Actual)

PRIMARY OUTCOMES:
postoperative pain intensity | 6 - 24 hours
  severity by visual analogue scale

SECONDARY OUTCOMES:
hospital stay | 1-5 days
  numbers of days

CONTACTS AND LOCATIONS:
Overall Officials: mohamed l ali, md, Study Director — Zagazig University
Locations (1):
- Zagazig University, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No